CLINICAL TRIAL: NCT03357484
Title: Influence of Leukocyte- and Platelet Rich Fibrin (L-PRF) on the Outcomes of Impacted Mandibular Third Molar Removal Surgery: a Split-mouth Randomized Clinical Trial
Brief Title: Leukocyte- and Platelet Rich Fibrin (L-PRF) Application in Impacted Mandibular Third Molar Removal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Povilas Daugela, DDS, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRF third molar
Record Dates: First submitted 2017-11-18; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Pain; Edema; Wound Heal
Keywords: impacted tooth; pain; platelet-rich fibrin; third molar; tooth extraction; wound healing
MeSH Terms: conditions — Pain; Edema; Tooth, Impacted | interventions — Leukocyte Count; Blood Coagulation

STUDY DESIGN:
Intervention Model Description: Patients who met the inclusion criteria for this split-mouth study underwent bilateral IMTM surgical extractions. Following extraction, randomization was done. One socket received L-PRF, and the other socket served as a regular blood clot control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and Independent Outcomes Assessor were blinded to study groups. Names of participants were coded and known to Principal investigator only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-PRF (Experimental): Third molar extraction sockets were filled with two leukocyte- and platelet rich fibrin (L-PRF) clots
  Interventions: Procedure: Leukocyte- and platelet rich fibrin
- Blood clot (Active Comparator): Third molar extraction sockets allowed to form a natural blood clot and undergo natural healing
  Interventions: Procedure: Blood clot

INTERVENTIONS:
Procedure: Leukocyte- and platelet rich fibrin — Prior to surgery, two 9 ml glass-coated tubes (Intra-Spin, Intra-Lock International, Boca Raton, USA) of patient venous blood were collected. Tubes were transferred to a centrifuge (Andreas Hettich GmbH & Co.KG, Tuttlingen, Germany) and processed for 12 minutes at 2800 rpm to prepare L-PRF.
  Arms: L-PRF
Procedure: Blood clot — Natural blood clot formed within extraction socket
  Arms: Blood clot

SUMMARY:
The purpose of this study was to evaluate the influence of leukocyte- and platelet-rich fibrin (L-PRF) on impacted mandibular third molar (IMTM) extraction wound healing, patient postoperative discomfort, and incidence of alveolar osteitis (AO).

Thirty patients (18 female, 12 male) who met the inclusion criteria for this split-mouth study underwent bilateral IMTM surgical extractions. Following extraction, randomization was done. One socket received L-PRF, and the other socket served as a regular blood clot control. Postoperatively, the soft tissue healing index (HI), pain according to visual analog scale (VAS), facial swelling using a horizontal and vertical guide, and incidence of AO were evaluated 1, 3, 7, and 14 days after surgery.

DETAILED DESCRIPTION:
The study was designed as a prospective split-mouth clinical trial on patients who needed bilateral paired IMTM extractions. The study was conducted at the Maxillofacial Surgery Department of the Lithuanian University of Health Sciences. Approval by the local bioethics committee was granted (No. BEC-MF-01). All patients signed an informed consent.

Patient selection Based on previously treated pilot cases, a power analysis was conducted for sample size estimation (Statistica 6.0, Dell Software, Round Rock, TX, USA). The calculations revealed a minimum sample size of n = 30, based on a power of 90% and an α of 5%.

The inclusion criteria were as follows:

1. Male and female patients with an age of 18 to 60 years;
2. Healthy patients (American Society of Anesthesiologists Physical Status (ASA PS) index ≤ 2);
3. Sole bilateral extractions of IMTMs during the same surgery;
4. Complete root formation of tooth No. 38 and 48 at radiological examination;
5. Absence of acute inflammation and/or infection in the IMTMs area;
6. No history of nonsteroidal anti-inflammatory drug (NSAID) use in the past 4 weeks prior to surgery;
7. Same-difficulty bilateral IMTM extractions, according to both Pederson and Juodzbalys & Daugela classifications;
8. Signed informed consent.

The following exclusion criteria were used:

1. Smoking patients;
2. IMTM surgery duration difference greater than 10 minutes for each side, seeking to avoid bias;
3. Different surgical manipulations taken at each IMTM surgery site;
4. Presence of any neoplastic lesion (benign or malignant), clinically or radiologically evaluable, at the site or close to the impacted tooth;
5. Presence of any radiolucent lesion >1 cm at impacted tooth level;
6. Absence of the adjacent tooth;
7. Systemic conditions or pharmacological treatments altering oral microbiota or immunologic response;
8. Alcohol or drug abuse;
9. Pregnant or breastfeeding women;
10. Lack of compliance by the patient or any other evidence suggesting that the patient was not likely to follow the study protocol.

Preoperatively, two blind expert surgeons assessed patient Orthopantomograph (OPG) and/or cone beam computed tomography (CBCT), evaluating IMTM extraction difficulty and complexity according to Pederson and Juodzbalys & Daugela indexes for each IMTM bilaterally. The overall kappa index for inter-observers agreement was calculated by using weighted kappa. Only teeth having the same extraction difficulty scores according to both classifications were enrolled in the study.

Pederson difficulty index assessment

Pederson difficulty index was evaluated based on anatomical and radiographic features of the tooth to be extracted. Following scores were given according to OPG and/or CBCT findings:

Spatial relationship

* Mesio angular 1
* Horizontal 2
* Vertical 3
* Distoangular 4

Depth

* Level A 1
* Level B 2
* Level C 3

Ramus relationship / space available

* Class I 1
* Class II 2
* Class III 3

According to the difficulty score total score, the IMTMs were classified as:

Minimally difficult (score 3 to 4) Moderately difficult (score 5 to 7) Very difficult (score 7 to 10).

Juodzbalys & Daugela classification Modification of the Juodzbalys & Daugela classification is related with the different interpretation of the final score, i.e. rating of surgical difficulty and the surgical time. Indexes and their evaluation remain unaltered. The impacted mandibular third molar is evaluated by considering its relationships with adjacent anatomical boundaries (second molar, mandibular ramus, alveolar crest, mandibular canal, corticals of the mandible) and its spatial position.

The classification attributes a score from ranging from 0 to 3 (0=conventional; 1=simple; 2=moderate; 3=complicated) to six items (M, R, A, C, B, S), according to the tooth positioning.

* in relation to the second molar (M): the wisdom tooth crown could be directed at, or above the equator of the second molar (conventional, score 0), directed below the equator, to the coronal third of the second molar root (simple, score 1), directed to the middle third of the second molar root (moderate, score 2), directed to the apical third of the second molar root (complicated, score 3)
* in relation to the mandibular ramus (R): the tooth could have sufficient space in the dental arch (conventional, score 0), could be partially impacted in the ramus (simple, score 1), completely impacted in the ramus (moderate, score 2), or completely impacted in the ramus in disto-angular or horizontal position (complicated, score 3).
* considering the apico-coronal position of the tooth in relationship with the alveolar crest (A): the tooth could be completely erupted (conventional, score 0), partially impacted but with the widest part of the crown (equator) above the bone (simple, score 1), partially impacted but the widest part of the crown below the bone (moderate, score 2), or completely encased into the bone (complicated, score 3).
* tooth relation with the mandibular canal is expressed as follows (C): ≥ 3 mm from the mandibular canal (conventional, score 0), contacting or penetrating the mandibular canal, with the wall of the mandibular canal which can be radiographically identified (simple, score 1), contacting or penetrating the mandibular canal, with the wall of the mandibular canal not radiographically identifiable (moderate, score 2), roots surrounding the mandibular canal (complicated, score 3).
* bucco-lingual position of the tooth in relation to mandibular lingual and buccal walls (B): closer to buccal wall (conventional, score 0), in the middle between lingual and buccal walls (simple, score 1), closer to lingual wall (moderate, score 2), closer to lingual wall, when the tooth is partially impacted or completely encased in the bone (complicated, score 3).
* the spatial tooth positioning (S) is defined as follows: vertical (conventional, score 0), mesio-angular at ≤ 60◦ (simple, score 1), disto-angular at ≥ 120◦ (moderate, score 2), horizontal or inverted (complicated, score 3).

L-PRF preparation Prior to surgery, two 9 ml glass-coated tubes (Intra-Spin, Intra-Lock International, Boca Raton, USA) of patient venous blood were collected. Tubes were transferred to a centrifuge (Andreas Hettich GmbH & Co.KG, Tuttlingen, Germany) and processed for 12 minutes at 2800 rpm to prepare L-PRF, as described previously.

Surgical procedure Surgical procedures were performed following a standardized surgical approach by one expert surgeon (PD). Surgical manipulations required for each tooth extraction were as follows: simple mobilization of the tooth, coronectomy, root separation, incision, osteotomy. After removal of IMTM and socket curettage, on the side randomly chosen by the opaque sealed envelope technique to be the study side, the extraction sockets were filled with two L-PRF clots, whereas on the other side (control), they were allowed to form a natural blood clot and undergo natural healing. Both sides were sutured with absorbable Polyglactin (Atramat, Internacional Farmacéutica S.A. de C.V., Mexico City, Mexico) interrupted 5-0 sutures. Patients were blinded to the study or control side selection.

Duration of the surgical procedure was counted from the beginning of surgical manipulations to complete removal of mandibular wisdom tooth and wound closure for each side separately. If there was a time difference greater than 10 minutes or if a different surgical manipulation was used between each bilateral extraction, the patient was excluded from the study.

Each patient was given systemic antibiotic prophylaxis (Clindamycin 600 mg per os) 1 hour before and 6 hours after surgery. Postoperatively oral Lornoxicam 8 mg was prescribed to use for pain control when needed. Patients were instructed to rinse with chlorhexidine 0.12% solution three times a day for 2 weeks and provided with both verbal and written postoperative instructions. The sutures were removed one week after surgery.

Postoperative outcome evaluation Quality of soft tissue healing, incidence of AO, pain, and facial swelling were selected as postoperative outcome measures.

Postextractional wound soft tissue healing evaluation Postextractional wound soft tissue healing was evaluated using a modified postextraction wound healing index (HI), which considered four parameters: bleeding, suppuration, tissue color, and consistency of the healing tissue. Each parameter involved 3 scoring levels; consequently, the cumulative scoring scale ranged from 4, corresponding to excellent healing, to 12, indicating severely impaired healing. HI was evaluated clinically by the same blinded examiner at the 1st, 3rd, 7th, and 14th days after surgery.

Alveolar osteitis evaluation Alveolar osteitis was characterized as postoperative continuous throbbing pain surrounding the alveolus that was not adequately relieved by analgesics and that increased in severity during a period of 1-3 days after tooth extraction. The pain was followed by partial or complete loss of the initial blood clot in the interior of the socket with or without halitosis.

Pain evaluation Pain was assessed using a written questionnaire with a visual analog scale (VAS) every day by the patient during the first postoperative week. VAS consisted of 10 units in combination with a graphic rating scale, where the leftmost score 0 represented absence of pain and the rightmost score 10 indicated the worst possible, unbearable, excruciating pain. Patients were blind to the knowledge of L-PRF and control sides and were asked to evaluate a VAS pain score for each operated side every day separately for the first week after surgery.

Facial swelling clinical assessment

Facial swelling clinical assessments were performed by a single blinded examiner at baseline (before surgery) and at the 1st-, 3rd-, and 7th-day visits postoperatively at approximately the same time of day. Patients were seated in a relaxed position with the inferior border of the mandible parallel to the floor. Facial swelling in the operation side was evaluated using two facial measurements with nonexpandable tape:

* In the vertical dimension, measurement from the lateral canthus of the eye to the pogonion of the mandible was taken;
* In the horizontal dimension, the distance from the lower border of the tragus to the mouth commissure on both operated sides was measured.

Facial swelling value was taken as the average value of these two measurements. The preoperative measurement was considered as the baseline value.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with an age of 18 to 60 years;
2. Healthy patients (American Society of Anesthesiologists Physical Status (ASA PS) index ≤ 2);
3. Sole bilateral extractions of IMTMs during the same surgery;
4. Complete root formation of tooth No. 38 and 48 at radiological examination;
5. Absence of acute inflammation and/or infection in the IMTMs area;
6. No history of nonsteroidal anti-inflammatory drug (NSAID) use in the past 4 weeks prior to surgery;
7. Same-difficulty bilateral IMTM extractions, according to both Pederson and Juodzbalys & Daugela classifications;
8. Signed informed consent.

Exclusion Criteria:

1. Smoking patients;
2. IMTM surgery duration difference greater than 10 minutes for each side, seeking to avoid bias;
3. Different surgical manipulations taken at each IMTM surgery site;
4. Presence of any neoplastic lesion (benign or malignant), clinically or radiologically evaluable, at the site or close to the impacted tooth;
5. Presence of any radiolucent lesion >1 cm at impacted tooth level;
6. Absence of the adjacent tooth;
7. Systemic conditions or pharmacological treatments altering oral microbiota or immunologic response;
8. Alcohol or drug abuse;
9. Pregnant or breastfeeding women;
10. Lack of compliance by the patient or any other evidence suggesting that the patient was not likely to follow the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain visual analogue scale (VAS) score change evaluation | 1st-, 2nd-, 3rd-, 4th-, 5th-, 6th-, and 7th- postoperative day
  Pain VAS scale consisted of 10 units in combination with a graphic rating scale, where the leftmost score 0 represented absence of pain and the rightmost score 10 indicated the worst possible, unbearable, excruciating pain.
Swelling change evaluation | 1st-, 3rd-, and 7th- postoperative day
  Facial swelling clinical assessments were performed by a single blinded examiner at baseline (before surgery) and at the 1st-, 3rd-, and 7th-day visits postoperatively at approximately the same time of day. Patients were seated in a relaxed position with the inferior border of the mandible parallel to the floor. Facial swelling in the operation side was evaluated using two facial measurements with nonexpandable tape:
  * In the vertical dimension, measurement from the lateral canthus of the eye to the pogonion of the mandible was taken;
  * In the horizontal dimension, the distance from the lower border of the tragus to the mouth commissure on both operated sides was measured.
  Facial swelling value was taken as the average value of these two measurements. The preoperative measurement was considered as the baseline value.
Healing index change evaluation | 1st-, 3rd-, 7th-, and 14th- postoperative day
  Postextractional wound soft tissue healing was evaluated using a modified postextraction wound healing index (HI) [24], which considered four parameters: bleeding, suppuration, tissue color, and consistency of the healing tissue. Each parameter involved 3 scoring levels; consequently, the cumulative scoring scale ranged from 4, corresponding to excellent healing, to 12, indicating severely impaired healing. HI was evaluated clinically by the same blinded examiner at the 1st-, 3rd-, 7th-, and 14th- after surgery.

OTHER OUTCOMES:
Alveolar osteitis | 2 postoperative weeks
  Alveolar osteitis was characterized as postoperative continuous throbbing pain surrounding the alveolus that was not adequately relieved by analgesics and that increased in severity during a period of 1-3 days after tooth extraction. The pain was followed by partial or complete loss of the initial blood clot in the interior of the socket with or without halitosis.

CONTACTS AND LOCATIONS:
Overall Officials: Povilas Daugela, DDS, Principal Investigator — Lithuanian University of Health Sciences; Vaidas Grimuta, DDS, Principal Investigator — Lithuanian University of Health Sciences; Dalius Sakavicius, DDS, PhD, Study Director — Lithuanian University of Health Sciences; Juozas Jonaitis, DDS, PhD, Principal Investigator — Lithuanian University of Health Sciences; Gintaras Juodzbalys, DDS, PhD, Study Chair — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No
There are no Plan to Share IPD